CLINICAL TRIAL: NCT06881121
Title: IMPLICATION OF FAST-TRACK PROTOCOL FOR HIP FRACTURE FIXATION IN ALEXANDRIA UNIVERSITY HOSPITALS: PROSPECTIVE CONTROLLED CLINICAL STUDY
Brief Title: IMPLICATION OF FAST-TRACK PROTOCOL FOR HIP FRACTURE FIXATION IN ALEXANDRIA UNIVERSITY HOSPITALS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Anas Ibrahim, Assistant lecturer Alexandria University, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMPLICATION OF FAST-TRACK
Record Dates: First submitted 2025-03-05; First posted 2025-03-18 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Fast-track Protocol; Hip Fracture; 30 Days Mortality
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Fast pathway (Experimental): Group Fast pathway: Seventy-five patients treated according to fast-track protocol.
  Interventions: Procedure: Fast-track protocol for hip fracture fixation
- Group Conventional pathway (No Intervention): Group Conventional pathway: Seventy-five patients who failed to be included in the fast track protocol will be included in the conventional (Non-Fast) pathway.

INTERVENTIONS:
Procedure: Fast-track protocol for hip fracture fixation — Fast-track protocol implication on mortality and morbidities in hip fracture fixation
  Arms: Group Fast pathway

SUMMARY:
The present study aims to evaluate the impact of fast-track protocol of hip fracture fixation within 48 hours on patients' mortality and morbidities. Primary aim is to observe the incidence of 30-day mortality of patients with hip fractures admitted to the operating room (OR) for fixation within 48 hours of the trauma event and to asses Deep vein thrombosis incidence, Pulmonary embolism incidence, Post-operative cognitive dysfunction, length of hospital stay.,Length of ICU stay,Patients who needed hospital readmission and the reasons and the success of the postoperative rehabilitation status.

DETAILED DESCRIPTION:
One hundred and fifty adult patients of American Society of Anesthesiologists (ASA) physical status I, II or III, age ≥ 50 years will be admitted to the department of orthopaedics surgery and traumatology, El Hadara University Hospital and scheduled for internal fixation under either spinal or general anaesthesia starting from January 2025. Patients will be divided into two groups: Group Fast pathway: Seventy-five patients treated according to fast-track protocol. Group Conventional pathway: Seventy-five patients who failed to be included in the fast track protocol will be included in the conventional (Non-Fast) pathway.

Preoperative evaluation and preparation: Evaluation of the patients will be carried out during the preoperative visit through proper history taking, clinical examination and routine laboratory investigations including complete blood picture, coagulation profile, blood urea, serum creatinine, serum electrolytes (sodium and potassium), fasting blood glucose, liver function tests and any other investigations needed. Serum lactate level informed written consent from all individual participants included in this study will be obtained during the preoperative visit. ECG, Echocardiograhy and Doppler lower limb examination for all patients. Fast-track care: The fast-track care will be started on admission to the hospital provided that the patients have fresh fractures. The patients will be examined in the emergency unit and directly transported to the radiology department with a tentative diagnosis of hip fracture. Preoperative treatment like administration of fascia iliaca compartment block (FICB) with a volume of 40 ml bupivacaine 0.25%, oxygen and prevention of pressure sores will be started. On arrival at the orthopaedic ward, standardised nursing routines (pain control, nutrition, fluid therapy and prevention of pressure sores) will begin. All patients with hip fracture will be scheduled for surgery within 48 hours. Whenever possible, all patients will be mobilised on the first postoperative day with a physiotherapist.

Specific comorbidities plan: Anaemia and blood transfusion: Packed RBCs transfusion will be ordered if preoperative Hb is < 8 gm/dL or 10 gm/dL in the presence of history of ischemic heart disease. Strategies to reduce blood loss include expediting surgery and minimising operating time, and the use of tranexamic acid. Cardiac condition assessment: An echocardiography will be ordered immediately, however surgery will not be delayed pending the results of echocardiography for undiagnosed ischemia; anaesthesia will instead proceed with invasive blood pressure monitoring and particular attention paid to maintaining cardiovascular stability through the use of lower doses of anaesthesia, i.v. fluids and vasoactive drugs as appropriate. Anti-platelets, anticoagulants and spinal anaesthesia: In case of the use of single antiplatelet therapy, including clopidogrel, spinal or general anesthesia will be allowed to proceed on a risk/benefit basis. (i) For patients taking vitamin K antagonists, spinal anaesthesia may be undertaken once the international normalised ratio (INR) is 1.5. Those patients presenting with an INR of >1.5 will receive an initial dose of vitamin K as soon as possible (i.e. in the emergency department), with further vitamin K or prothrombin complex concentrate if the INR remains >1.5 after 4-6 h. Bridging therapy (e.g. heparin infusion) will be ordered for complex patients like those with a metallic heart valve. (ii) For patients with direct-acting oral anticoagulant (DOAC), spinal or general anaesthesia will be allowed after two half-lives have elapsed. CKD patients: If creatinine > 2 mg/dl, this will need additional precautions:

- Potentially nephrotoxic drugs will be stopped e.g. NSAIDs, ACEI, diuretics. - Good hydration will be ensured. - Patients will be catheterised and a fluid balance chart will be started. Surgery will be allowed to proceed after ensuring good urine output. All patients who failed to be included in the fast track protocol (non-fast track) will be managed accordingly and followed, and the results will be compared to the fast track group. Pre-anaesthetic preparation and premedication: Fasting hours (6 hours to solids and 2 hours to clear fluids). Thrombotic prophylaxis (enoxaparin 40 mg) will be started 12 hours before surgery unless on bridging therapy. Antiseptic shower will be provided. Antibiotic prophylaxis: single dose ceftriaxone 2 g intravenously will be given 1 hour before surgical incision according to the hospital policy. Fluids and nutrition: Intravenous fluid (Ringer's) administered at a rate of 1 litre over 8 hours or according to renal and cardiac recommendations. A resuscitation fluid bolus of 5-10 ml/kg will be considered. On arrival to the operative theatre: A peripheral cannula (18G) will be inserted to all patients. A multichannel monitor (Dräger® Infinity vista XL) will be connected to the patient to display continuous electrocardiography monitoring for heart rate (beat/min) and rhythm, noninvasive arterial blood pressure (NIBP), arterial oxygen saturation (SpO2) and end-tidal carbon dioxide (ETCO2).

Anaesthesia: Patients will receive either spinal or general anaesthesia with FICB. Patients will be given spinal anesthesia with a maximum dose of 2.5 ml 0.5% hyperbaric bupivacaine at the L3/4 interspaces (alternatively at the L2/3 or L4/5 interspaces) under complete aseptic technique. If the patient has contraindication to spinal anaesthesia, general anaesthesia will be conducted. General Anaesthesia: preoxygenation for 3 minutes, standard anaesthesia will be induced with propofol in increments up to 2mg/kg till loss of verbal response, fentanyl 1μg/kg and atracurium 0.5 mg/kg intravenously to facilitate tracheal intubation or laryngeal mask airway (LMA) insertion. Anaesthesia will be maintained with 50% oxygen in air and isoflurane 1-1.5 MAC to maintain adequate depth of anaesthesia. The haemodynamic variables (eg, heart rate or blood pressure) will be maintained within 20% of the preoperative baseline values and if not, patients will be treated with additional boluses of fentanyl 0.5 mcg/kg intraoperatively as needed. Mechanical ventilation will be performed with a constant tidal volume of 6-8 ml/ kg and a respiratory rate of 10 to 12 cycles/min to maintain the end-tidal carbon dioxide tension between 35 and 40 mmHg and an oxygen saturation of ≥ 98 % with 50 % oxygen in air. Incremental doses of atracurium 0.1 mg/kg will be administered to maintain muscle relaxation according to nerve stimulator. The FICB: After spinal or general anaesthesia, the patient will be placed in complete supine position with the legs extended flattened to maximize access to the inguinal area, although palpation of a femoral pulse is a useful landmark, it is not required because the artery is quickly visualized by placement of the transducer transversely on the inguinal crease, followed by slow movement laterally or medially. Tilting the probe while pressing helps to identify the hyperechoic fascia iliaca superficial to the hypoechoic iliopsoas muscle. Medially, the femoral nerve is visualized deep to the fascia and lateral to the artery. Laterally, the sartorius muscle is identified by its typical triangular shape when compressed by the transducer. The goal is to place the needle tip under the fascia iliaca approximately at a lateral third of the line connecting the anterior superior iliac spine to the pubic tubercle (the injection is made several centimeters lateral to the femoral artery) and to deposit a volume of 40 ml bupivacaine 0.25%. A proper injection will result in the separation of the fascia iliaca by the local anaesthetic in the medial-lateral direction from the point of injection as described. In both types of Anaesthesia: if the MAP drops below 60 mmHg, ephedrine 10 mg IV bolus and fluid bolus will be given and repeated if required. Atropine 0.5 mg IV bolus will be given if HR decreases to less than 50 beats/min. Normothermia will be maintained using bair hugger and warm intravenous fluids. Urinary catheter will be inserted for monitoring of urine output. All the procedures will be performed by expert surgeons with a clinical experience of more than 5 years. At the end of surgery, anaesthesia will be discontinued; residual neuromuscular block will be reversed by atropine 0.02 mg/kg and neostigmine 0.025 - 0.05 mg/kg. Extubation will be performed awake after the return of protective airway reflexes. Anti-emetic measures: ondansetron 8 mg intravenously will be administered at the end of surgery. Postoperative Management: All patients will be transferred to the intermediate care unit and will be closely monitored continuously for the next 24 hours. Multimodal analgesia in the form of intravenous paracetamol 1 g/8 hours (Perfalgan® 100 ml vial UPSA France) and intravenous ketorolac 15 mg/8 hours will be administered for postoperative pain control. If the VAS score is ≥ 4, FICB will be reconsidered with 40 ml 0.1 % bupivacaine. The incidence of postoperative nausea and vomiting (PONV) will be assessed by a nurse for the first 24 hours and only 2 possible answers will be accepted (yes or no). Nausea is defined as subjective sensation of discomfort associated with the awareness of the urge to vomit. Vomiting is defined as a forceful expulsion of gastric contents through the mouth.Rescue antiemetic ondansetron 8 mg intravenously will be given if the patient has persistent nausea or more than a single episode of vomiting. Removal of urinary catheter will be encouraged as early as possible after surgery. DVT prophylaxis: LMWH will be continued postoperatively no earlier than 4 hours after the procedure. Rehabilitation: Physiotherapy assessment and early mobilisation of all patients the day following surgery will be done. Nutrition management: multidisciplinary team including orthogeriatricians, occupational therapists and nutritionists will be organized for optimization of nutrition state. Combined oral and parenteral supplementation will be ordered to increase the daily nutritional intake to near-optimum levels (nutrition levels based on basal demand of 25 kcal/kg body weight/day and fluid levels based on 30 mL/kg body weight/day) or according to renal and cardiac recommendations.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50 years.
2. ASA physical status class I, II or III.

Exclusion Criteria:

1. Poly-trauma patients.
2. Patients with history of sensitivity to the studied drugs.
3. Psychiatric disease or seizure disorder requiring medication within the previous 2 years.
4. Opioid tolerant patients.
5. Patients with preoperative cognitive dysfunction.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
30 days mortality | 30 days post operative
  Mortality: The follow-up time will be 30 days either through postoperative visits or phone call and documented. Time to death will be calculated from admission to possible event.

SECONDARY OUTCOMES:
Time to surgery | Hours before surgery
  Time to surgery (TTS) will be calculated as hours from fracture time to surgery.
Duration of surgery | During Surgery
  Duration of surgery (mins).
Deep vein thrombosis incidence | Post opertaive day 5
  Any patient with suspected signs of DVT postoperatively will be confirmed with a doppler examination and documented.
Pulmonary embolism incidence | Post operative day 5
  The diagnosis of pulmonary embolism if suspected clinically by Wells' criteria will be confirmed with pulmonary angiography, transferred to ICU and managed accordingly.
Thromboembolic complications | Post opertaive day 5
  Thromboembolic complications: as stroke and MI will be confirmed by CT brain and cardiac enzymes and transferred to ICU and managed accordingly.
Length of ICU stay | Post opertaive day 5
  Length of ICU stay (days): The numbers of days from ICU admission to discharge.
Length of hospital stay | Post opertaive day 5
  Length of hospital stay (days): LOS is defined as the number of days between the operation and discharge from the hospital.
Cause of delay in non-fast track protocol. | Perioperative
  Cause of delay in non-fast track protocol.
Cognitive dysfunction | T0: during preoperative visit. T1: 120 minutes postoperatively. T2: 24 hours postoperatively.
  Cognitive dysfunction using Mini Mental State Examination (MMSE) test will be recorded
Incidence of postoperative nausea and vomiting | 24 hours post operative
  Incidence of postoperative nausea and vomiting in the first 24 hours postoperatively.
Number of patients requiring rescue anti-emetic | 24 hours post operative
  Number of patients requiring rescue anti-emetic postoperatively will be recorded.
Incidence of infection and complications | Post opertaive day 5
  Incidence of infection and complications: as chest infection, UTI and surgically related infections.
Serum lactate level (mmol/L) | 12 hours preoperative and 24 hours post operative
  Serum lactate level (mmol/L): will be measured preoperatively and 12 hours postoperatively for detection of possible hypoperfusion.
Patients who needed hospital readmission | Up to 30 days postoperative
  Patients who needed hospital readmission and the reasons.
The reasons of hospital readmission | Up to 30 days postoperative
  The reasons of hospital readmission
Rehabilitation status | Up to 30 days postoperative
  Rehabilitation status will be assessed during the 30 day postoperative follow up period: the following will be assessed during postoperative visit - Patients who walked assisted. - Patients who continued to need nursing home care.

CONTACTS AND LOCATIONS:
Overall Officials: Moustafa Abdelaziz Ahmed, MD, Study Director — Alexandria University; Maher Doghiem, MD, Study Director — Alexandria University; Ahmed Shehab, MD, Study Director — Alexandria University
Locations (1):
- Faculty of medicine Alexandria University, Alexandria, Egypt, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Throug clinical trials
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2 years
Access Criteria: Fast-track Hip fracture fixation